CLINICAL TRIAL: NCT01920698
Title: Multicentre Randomized Study of Percutaneous Mitral Valve Repair MitraClip Device in Patients With Severe Secondary Mitral Regurgitation.
Brief Title: Multicentre Study of Percutaneous Mitral Valve Repair MitraClip Device in Patients With Severe Secondary Mitral Regurgitation
Acronym: MITRA-FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013.798; 2013-A00464-41 (Other: IDRCB)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: Heart Valve Diseases; Heart failure; Heart diseases; Mitral valve insufficiency
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases; Heart Failure; Heart Diseases; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MitraClip Device (Experimental): Subjects randomized to the MitraClip Device group will undergo the MitraClip procedure in addition to optimal standard medical therapy.
  Interventions: Device: Percutaneous MitraClip Device Implantation
- Control (Other): Patients randomized to the Control group will receive optimal therapy alone
  Interventions: Other: control

INTERVENTIONS:
Device: Percutaneous MitraClip Device Implantation — MitraClip System includes a MitraClip device, a steerable guide catheter and a MitraClip delivery system
  Arms: MitraClip Device
Other: control
  Other Names: Patients randomized to the Control Group will receive optimal medical therapy alone
  Arms: Control

SUMMARY:
The objective of this trial is to compare the safety, the efficacy and the cost-effectiveness of 2 therapeutic strategies (optimal standard of care therapy alone versus percutaneous MitraClip procedure and optimal standard of care therapy) in patients with severe secondary mitral regurgitation.

This trial is a French, multicenter and randomized trial. Patients enrolled will be clinically followed for 2 years (phone call at 1 month, clinical visit at 6 months, 12 months and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Severe secondary mitral regurgitation characterised, according to the European guidelines and recommendations, by a regurgitant volume>30 mL/beat or an effective regurgitant orifice>20 mm².
* New York heart Association Class≥ II.
* Left ventricular ejection fraction between 15% and 40%
* Minimum of 1 hospitalization for heart failure within 12 months preceding randomization
* Optimal standard of care therapy for heart failure according to investigator.
* Not eligible for a mitral surgery intervention according to the Heart Team.
* Willingness to participate in the study and signed written informed consent
* Affiliation to a health insurance system or a similar system

Exclusion Criteria:

* Eligible for a mitral surgery intervention according to the Heart Team.
* Primary mitral regurgitation.
* Myocardial infarction or coronary bypass grafting surgery within three months prior to randomization.
* Cardiac resynchronization therapy within three months prior to randomization.
* Cardioversion within three months prior to randomization
* Transcatheter aortic valve implantation within three months prior to randomization
* Need for any cardiovascular surgery (including registration on cardiac transplant list).
* Coronary angioplasty within one month prior to randomization.
* Previous surgical mitral valve repair.
* Renal replacement therapy.
* Active infection requiring current antibiotic therapy.
* Severe hepatic insufficiency.
* Stroke within three months prior to randomization.
* Concurrent medical condition with a life expectancy of less than 12 months.
* Uncontrolled arterial hypertension.
* Hypersensitivity to nitinol.
* Participation to another trial.
* Pregnancy.
* No affiliation to a health insurance system.
* Legal protection measure (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and unplanned hospitalizations for heart failure | 1 year

SECONDARY OUTCOMES:
All-cause mortality, cardiac mortality | 30 days, 6 months, 12 months, and 24 months.
Survival with no major cardiovascular events | 30 days, 6 months, 12 months, and 24 months.
Serious Adverse Events | 30 days, 6 months, 12 months and 24 months.
  Any serious adverse events cardiovascular or not occurring within each group.
Change in Quality of Life score as measured by the European Quality of Life-5 Dimensions instrument. | 6 months and 12 months
Change in functional evaluation | 12 months
Change in echocardiographic evaluation between baseline at 6, 12 and 24 months. | 6 months, 12 months and 24 months
Change in biomarkers (BNP levels, creatinine) at 6 months and 12 months | 6 months and 12 months
Cost-effectiveness of each strategy at 12 months | 12 months
  Cost-effectiveness of each therapeutic strategy will be assessed by the evaluation of medical costs linked to the pathology (hospitalizations, consultations, and external medical costs (biology, radiology, medications) and compared in the 2 groups during the first 12 months of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: JEAN FRANCOIS OBADIA, MD, Principal Investigator — Hospices Civils de Lyon
Locations (40):
- France (40):
  - CHU d'Angers, Angers
  - Chu de Besancon, Besançon
  - Chu de Bordeaux, Bordeaux
  - CHRU La Cavale Blanche, Brest
  - Groupement Hospitalier Est, Bron
  - CHU Caen, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - APHP Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital privé de Parly 2, Le Chesnay
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Chu de Lille, Lille
  - Hôpital privé le Bois, Lille
  - Hôpital Saint-Joseph, Marseille
  - Hopital de La Timone, Marseille
  - Hôpital privé Clairval, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - CH Annecy Genevois, Metz-Tessy
  - Chu de Montpellier, Montpellier
  - Clinique Du Millenaire, Montpellier
  - Chu de Nancy, Nancy
  - Chu de Nantes, Nantes
  - Centre chirurgicale Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Pasteur, Nice
  - Groupe Hospitalier La Salpétrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Aphp Hopital Bichat, Paris
  - CHRU La Milétrie, Poitiers
  - Chu de Rennes, Rennes
  - CHU Rouen, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Hôpital Nord, Saint-Etienne
  - Institut Arnault Tzanck, Saint-Laurent-du-Var
  - Chu de Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - Chu de Toulouse, Toulouse
  - CHRU de Tours, Tours
  - Clinique Cardiologique Saint Gatien, Tours
  - Clinique du Tonkin, Villeurbanne

REFERENCES:
- [Background] Obadia JF, Armoiry X, Iung B, Lefevre T, Mewton N, Messika-Zeitoun D, Cormier B, Berthiller J, Maucort-Boulch D, Boutitie F, Vaz B, Trochu JN, Vahanian A. The MITRA-FR study: design and rationale of a randomised study of percutaneous mitral valve repair compared with optimal medical management alone for severe secondary mitral regurgitation. EuroIntervention. 2015 Mar;10(11):1354-60. doi: 10.4244/EIJV10I11A232. PMID 25798568
- [Background] Iung B, Armoiry X, Vahanian A, Boutitie F, Mewton N, Trochu JN, Lefevre T, Messika-Zeitoun D, Guerin P, Cormier B, Brochet E, Thibault H, Himbert D, Thivolet S, Leurent G, Bonnet G, Donal E, Piriou N, Piot C, Habib G, Rouleau F, Carrie D, Nejjari M, Ohlmann P, Saint Etienne C, Leroux L, Gilard M, Samson G, Rioufol G, Maucort-Boulch D, Obadia JF; MITRA-FR Investigators. Percutaneous repair or medical treatment for secondary mitral regurgitation: outcomes at 2 years. Eur J Heart Fail. 2019 Dec;21(12):1619-1627. doi: 10.1002/ejhf.1616. Epub 2019 Nov 18. PMID 31476260
- [Result] Obadia JF, Messika-Zeitoun D, Leurent G, Iung B, Bonnet G, Piriou N, Lefevre T, Piot C, Rouleau F, Carrie D, Nejjari M, Ohlmann P, Leclercq F, Saint Etienne C, Teiger E, Leroux L, Karam N, Michel N, Gilard M, Donal E, Trochu JN, Cormier B, Armoiry X, Boutitie F, Maucort-Boulch D, Barnel C, Samson G, Guerin P, Vahanian A, Mewton N; MITRA-FR Investigators. Percutaneous Repair or Medical Treatment for Secondary Mitral Regurgitation. N Engl J Med. 2018 Dec 13;379(24):2297-2306. doi: 10.1056/NEJMoa1805374. Epub 2018 Aug 27. PMID 30145927
- [Derived] Iung B, Messika-Zeitoun D, Boutitie F, Trochu JN, Armoiry X, Maucort-Boulch D, Obadia JF, Vahanian A. Characteristics and Outcome of COAPT-Eligible Patients in the MITRA-FR Trial. Circulation. 2020 Dec 22;142(25):2482-2484. doi: 10.1161/CIRCULATIONAHA.120.049743. Epub 2020 Dec 21. No abstract available. PMID 33347327
- [Derived] Messika-Zeitoun D, Iung B, Armoiry X, Trochu JN, Donal E, Habib G, Brochet E, Thibault H, Piriou N, Cormier B, Tribouilloy C, Guerin P, Lefevre T, Maucort-Boulch D, Vahanian A, Boutitie F, Obadia JF. Impact of Mitral Regurgitation Severity and Left Ventricular Remodeling on Outcome After MitraClip Implantation: Results From the Mitra-FR Trial. JACC Cardiovasc Imaging. 2021 Apr;14(4):742-752. doi: 10.1016/j.jcmg.2020.07.021. Epub 2020 Sep 16. PMID 32950444